CLINICAL TRIAL: NCT05200208
Title: Improving Sleep and Cognition in Alzheimer's Disease: A Pilot RCT of Citicoline
Brief Title: Improving Sleep and Cognition in Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Emory Goizueta Alzheimer's Disease Research Center (ADRC) (Unknown)
Responsible Party: Principal Investigator, Victoria Pak, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002909; P50AG025688 (NIH); 2025P010359 (Other: Emory IRB)
Record Dates: First submitted 2022-01-18; First posted 2022-01-20 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease
Keywords: Sleep disturbance
MeSH Terms: conditions — Alzheimer Disease; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Citicoline Supplement (Experimental): Participants with AD will receive a dietary citicoline supplement
  Interventions: Dietary Supplement: Citicoline supplement
- Placebo (Placebo Comparator): Participants with AD will receive a placebo supplement
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Citicoline supplement — Participants with AD will receive a dietary citicoline supplement. Subjective sleep measures will be measured via the Pittsburgh Sleep Quality Index (for measurement of sleep quality) and Epworth Sleepiness Scale (for measurement of sleepiness). Cognition will be measured by Rey Auditory Verbal Learning Test (RAVLT), Trail Making Test (TMT) Parts A & B, and the Montreal Cognitive Assessment (MOCA). Participants will complete all questionnaires at baseline and at follow-up at 3 months.
  Arms: Citicoline Supplement
Other: Placebo — Participants with AD will receive a placebo supplement. Subjective sleep measures will be measured via the Pittsburgh Sleep Quality Index (for measurement of sleep quality) and Epworth Sleepiness Scale (for measurement of sleepiness). Cognition will be measured by Rey Auditory Verbal Learning Test (RAVLT), Trail Making Test (TMT) Parts A & B, and the Montreal Cognitive Assessment (MOCA). Participants will complete all questionnaires at baseline and at follow-up at 3 months.
  Arms: Placebo

SUMMARY:
Cognitive disorders include such things as memory disorders, mild cognitive impairment, and Alzheimer's disease (AD). The purpose of the study is to learn more about whether a dietary citicoline supplement will improve sleep and cognition. Sleep disturbances currently afflict approximately 25-44% of those with AD, resulting in decreased quality of life for those with AD and their caregivers and are a major driver of institutionalization.

Previous studies have tested this dietary supplement in Alzheimer's disease and shown that citicoline may improve cognitive decline. The research team would like to see if citicoline will also improve sleep. The citicoline that will be provided is made by Kyowa Hakko Pharma Chemical Company. This dietary supplement has been tested for Alzheimer's disease and found to be well tolerated. Citicoline has previously been used safely in other Alzheimer's disease populations at the same dosage.

DETAILED DESCRIPTION:
The research team will test these hypotheses via a randomized, double-blind, placebo-controlled pilot study of citicoline in individuals with AD. Participants will be recruited from the Alzheimer's Disease Research Center (ADRC) and from the community in the surrounding Atlanta area. This will be a 3-month randomized, double-blind, placebo-controlled trial comparing citicoline and placebo in a well-characterized cohort of 20 individuals with AD. Subjective sleep measures will be measured via the Pittsburgh Sleep Quality Index (for measurement of sleep quality) and Epworth Sleepiness Scale (for measurement of sleepiness). For neuropsychological and cognition will be measured measures, the research team will employ the Rey Auditory Verbal Learning Test (RAVLT), Trail Making Test (TMT) Parts A & B, and the Montreal Cognitive Assessment (MOCA).

Those participating in the ADRC parent study or recruited from the community and diagnosed with AD in their medical record and aged 18 and over are eligible to participate. Eligible participants will be enrolled in a two-treatment trial comparing the effects of citicoline (1000 mg once per day with or without food) to a placebo. There will be a baseline (T0) visit and a follow-up 3 months later (T1) as a separate visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are diagnosed with AD and confirmed from the medical record.
* At least 18 years of age living within the continental United States
* Read and understand English
* Have Internet and email access (this criterion applies to the legally authorized representatives)

Exclusion Criteria:

* No telephone access
* Epilepsy or head trauma resulting in unconsciousness in the past two years
* Presence of chronic obstructive pulmonary disease, asthma, severe cardiac insufficiency (congestive heart failure, myocardial infarction), type I diabetes, vitamin B12 or folic acid deficiency, liver cirrhosis, thyroid dysfunction, rheumatoid arthritis, chronic renal failure, and/or psychiatric disorders, obstructive sleep apnea, restless legs syndrome or periodic limb movement disorder
* History of alcohol dependence and medication abuse
* Night shift workers or those in situations where they regularly experience jet lag, or have irregular work schedules, since circadian misalignment may alter markers of inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2025-09-21 (Actual); Study Completion 2025-09-21 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Baseline and 3 months
  Impact on sleep by the administration of the citicoline supplement will be assessed by completing the Pittsburgh Sleep Quality Index (PSQI): This questionnaire is used to measure subjective sleep quality. It has strong validity and reliability in clinical populations and consists of 19 items asking about sleep disturbances over the past month with 7 dimensions. Each dimension scores 0 (no difficulty) to 3 (severe difficulty) and the sum of these scores yields a global sleep quality score that ranges from 0-21. Higher scores indicate greater difficulty sleeping. This questionnaire can be filled out by the participant, caregiver, or both as appropriate.
Epworth Sleepiness Scale (ESS) Change in the impact on daytime sleepiness by the administration of the citicoline supplement. | Baseline and 3 months
  The impact on daytime sleepiness will be assessed by completing the Epworth Sleepiness Scale (ESS). The ESS is a clinical and research standard used to determine perceived daytime sleepiness over the past month. It is a self-administered, validated questionnaire and takes approximately 2-3 minutes to complete. Respondents are asked to rate how likely they are to doze off in 8 situations, from 0 (would never doze) to 3 (high chance of dozing). Any score of 10 or above is considered an indicator of pathologic sleepiness. This questionnaire can be completed by the participant, caregiver, or both as appropriate.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Baseline and 3 months
  To examine how a change in sleep correlates with changes in cognitive function following the administration of citicoline, an assessment of cognitive function will be performed using the Montreal Cognitive Assessment (MoCA). The MoCA assesses global cognitive function and is a rapid screening instrument that takes approximately 10 minutes. It assesses various cognitive domains, including attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. This questionnaire will be administered to the participant through the ADRC at their baseline visit, and the researchers will measure it separately at their follow-up visit at 3 months. The total is out of 30 points. Scores below 26 can suggest varying degrees of cognitive impairment. For example, scores between 18 and 25 may indicate mild impairment, while scores between 10 and 17 might suggest moderate impairment.
Rey Auditory Verbal Learning Test (RAVLT) | Baseline and 3 months
  To examine how a change in sleep correlates with changes in memory function with the administration of citicoline,the research team will use the Rey Auditory Verbal Learning Test (RAVLT): RAVLT evaluates the nature and severity of memory dysfunction and is used to track changes in memory function in patients over time. It is designed to present a list of 15 words across five consecutive trials. The list is first read aloud to the participant, and the participant is immediately asked to recall as many words as possible.
Trail Making Test (TMT) | Baseline and 3 months
  To examine how a change in sleep correlates with changes in executive functioning with the administration of citicoline, participants will complete the Trail Making Test (TMT) Parts A & B: TMT assesses executive functioning. The test consists of two parts-Part A and Part B. In Part A, participants are asked to draw lines sequentially connecting 25 numbers distributed on paper. In Part B, in contrast, participants are asked to draw lines sequentially, while alternating between numbers and letters. The time spent to complete the task will be recorded for evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Pak, PhD, MS, MTR, Principal Investigator — Emory School of Nursing, School of Public Health
Locations (2):
- United States (2):
  - Emory University School of Nursing, Atlanta, Georgia
  - Goizueta Alzheimer's Disease Research Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT05200208/ICF_000.pdf